CLINICAL TRIAL: NCT05716373
Title: The Effect of Reiki Application on Pain, Fatigue and Sleep Quality in Elderly Persons Staying in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gülcan Bahçecioğlu Turan, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-97132852-050.01.04-162832
Record Dates: First submitted 2023-01-28; First posted 2023-02-08 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Pain; Tiredness; Sleep Quality
MeSH Terms: conditions — Pain; Fatigue; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: reiki
Who Masked: Participant
Masking Description: Single (Participant) pain,tiredness,sleep quality
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: (Experimental): reiki will be aplicated
  Interventions: Behavioral: pain
- control (No Intervention): Routine maintenance will be applied.

INTERVENTIONS:
Behavioral: pain — reiki
  Other Names: tiredness; sleep quality
  Arms: Experimental:

SUMMARY:
A person's life is a stage that passes in the time interval that ends with his birth when he opens his eyes to the world and his death when he closes his eyes to the world. Old age is a forced end for all people. Sleep is one of the most important and basic human needs. It prepares the individual for a new day by resting the body, strengthening and regulating the cerebral functions and repairing the brain. While a change in sleep pattern and quality affects a person's daily life activities, long-term persistence of this change may lead to deterioration of body and mental health.During Reiki practices, the hands are held in each position for 3-5 minutes by touching the head, neck, chest, abdominal cavity and groin. In problem areas, this time can be extended to 10-20 minutes. The duration of treatment lasts an average of 30-90 minutes. During the application, the person is in a lying or lying position and does not need to take off his clothes.

DETAILED DESCRIPTION:
In the elderly, the pathology of fatigue has not yet been fully elucidated. Natural changes and the disadvantages of age can be the cause of fatigue. Decrease in muscle strength, sarcopenia, pain, inactivity, changes in body composition due to malnutrition, decrease in physical fitness, insufficient energy systems, cardiovascular and respiratory problems, medications used can cause fatigue in the elderly. It has been shown that 27-50% of the elderly suffer from moderate to severe fatigue. Increasing the severity of fatigue reduces the daily activity performance of the elderly (6). Today, in many areas, in addition to medical treatment to reduce the symptoms of chronic diseases, alternative and complementary medicine are also used. Reiki, which constitutes our research subject; one of the energy approaches, in Japan at the end of the 19th century, Dr. It is a complementary medicine application discovered by Usui in Sanskrit inscriptions, which has been shown to be effective on pain, depression, insomnia and fatigue symptoms. Reiki is generally safe and no serious side effects have been reported. Reiki practice in the last 10 years; it increases among physicians, nurses and other health workers.

ELIGIBILITY:
Inclusion Criteria:

* • Being a nursing home resident and being 50 years or older,

  * Not having a communication problem,
  * Not having been diagnosed with bipolar disorder, schizophrenia or other mental illness,
  * Not taking antidepressant treatment,
  * Having chronic pain (arthralgia, back pain, musculoskeletal pain - at least once a day),
  * Not using a pain reliever all the time,
  * Willingness to participate in a four-week reiki program,
  * Not having received body-mind therapy (yoga, reiki, massage, meditation) in the last six months.
  * Having a scale score of >5 on the Piper Fatigue Scale
  * A score of >5 on the Pittsburgh Sleep Quality Scale
  * A scale score of >5 on the Visual Analog Scale

Exclusion Criteria:

* Needing antidepressant treatment,
* Not getting bored with work and not wanting to answer questions.

Exclusion Criteria:

-

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PUKI); | 1 hours later
  The scale is a safe and consistent questionnaire that evaluates the amount of sleep, sleep quality, presence and severity of sleep disorders in individuals in the last month.There are seven components in PUKI. These components are subjective sleep quality (component 1), sleep latency (component 2), sleep duration (component 3), habitual sleep efficiency (component 4), sleep disturbance (component 5), sleep medication use (component 6) and daytime dysfunction. (component 7). The evaluation score of each item is between 0-3. The total score obtained varies between 0-21. The higher the score, the worse the sleep quality. A score greater than five indicates poor sleep quality.
Piper Fatigue Scale | 1 hours later
  The scale evaluates the individual's subjective perception of fatigue in four sub-dimensions. These; behavior/violence sub-dimension evaluating the effect and severity of fatigue on activities of daily living (ADLs (6 items; 2-7); affect sub-dimension, which includes the emotional meaning attributed to fatigue (5 items; 8-12); it is the sensory sub-dimension (5 items; 13-17) that reflects the mental, physical and emotional symptoms of fatigue, and the cognitive/spiritual sub-dimension that reflects the effect of fatigue on cognitive functions and mental state (6 items; 18-23). As a result of the average score; 0 points are interpreted as no fatigue, 1-3 points as mild fatigue, 4-6 points as moderate fatigue, 7-10 points as severe fatigue. High scores obtained from the scale mean that the perceived fatigue level is high.
Visual Analog Scale (VAS) Evaluation | 1 hours later
  The Visual Analog Scale (VAS) is used to convert some values that cannot be measured numerically. Two end definitions of the parameter to be evaluated are written at the two ends of a 100 mm line, and the patient is asked to indicate where on this line their situation is appropriate by drawing a line or by placing a dot or pointing. For example, for pain, I have no pain at one end and very severe pain at the other end and the patient marks his/her current state on this line. The length of the distance from the point where there is no pain to the point marked by the patient indicates the patient's pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Gülcan B Turan, Elâzığ, Merkez, Turkey (Türkiye)